CLINICAL TRIAL: NCT03560089
Title: Serious Games Rehabilitation Programme to Treat Gant and Balance Disorders in Patients With Parkinson's Disease
Brief Title: Serious Games Rehabilitation Programme to Treat Gait and Balance Disorders in PD Patients
Acronym: PARKGAME-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C17-07
Record Dates: First submitted 2018-05-15; First posted 2018-06-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Gait; Rehabilitation; Serious game
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded assessment of video
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation with active serious game (Active Comparator): 25 patients will perform motor rehabilitation programme using the serious game
  Interventions: Device: Serious game
- No active serious game (Placebo Comparator): 25 patients will not perform motor rehabilitation programme using the serious game
  Interventions: Device: Placebo serious game

INTERVENTIONS:
Device: Serious game — Serious game with movements
  Arms: Rehabilitation with active serious game
Device: Placebo serious game — Serious game without movement
  Arms: No active serious game

SUMMARY:
To test the effects of a serious game rehabilitation programme in 50 patients with Parkinson's disease with gait and balance disorders in a randomised controlled study

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Gait and balance disorders resistant to dopaminergic medication

Exclusion Criteria:

* dementia
* contra-indication to magnetic resonance imaging

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Duration of the time-up-go test | change between baseline and at 6 weeks

SECONDARY OUTCOMES:
Duration of the time-up-go test | change between baseline and at 18 weeks
Step length | change between baseline and at 6 weeks
step velocity | change between baseline and at 6 weeks
Movement disorders Unified Parkinson's disease rating scale | change between baseline and at 6 weeks
freezing of gait questionnaire | change between baseline and at 6 weeks
Parkinson's disease quality of life scale | change between baseline and at 6 weeks
gait and balance scale | change between baseline and at 6 weeks
Montreal Cognitive Assessment | change between baseline and at 6 weeks
Magnetic resonance imaging | change between baseline and at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marie Laure Welter, PH MD PHD, Principal Investigator — ICM, 47 bd de l'Hôpital, 75013 Paris
Locations (1):
- Centre Investigation Clinique- ICM, Paris, France

REFERENCES:
- [Background] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Result] Skrzatek A, Nuic D, Cherif S, Beranger B, Gallea C, Bardinet E, Welter ML. Brain modulation after exergaming training in advanced forms of Parkinson's disease: a randomized controlled study. J Neuroeng Rehabil. 2024 Aug 5;21(1):133. doi: 10.1186/s12984-024-01430-w. PMID 39103924
- [Result] Nuic D, van de Weijer S, Cherif S, Skrzatek A, Zeeboer E, Olivier C, Corvol JC, Foulon P, Pastor JZ, Mercier G, Lau B, Bloem BR, De Vries NM, Welter ML. Home-based exergaming to treat gait and balance disorders in patients with Parkinson's disease: A phase II randomized controlled trial. Eur J Neurol. 2024 Jan;31(1):e16055. doi: 10.1111/ene.16055. Epub 2023 Sep 10. PMID 37691341
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886